CLINICAL TRIAL: NCT05272332
Title: Serial Ultrasound Assessment of Gastric Volume in Mechanically Ventilated Patients Fasted Prior to Extubation: a Prospective Observational Study
Brief Title: Gastric Ultrasound Prior to Extubation
Status: Completed | Type: Observational
Sponsor: Prince of Wales Hospital, Shatin, Hong Kong (Other)
Responsible Party: Principal Investigator, Esther Tang, Principle Investigator, Prince of Wales Hospital, Shatin, Hong Kong
Other Study IDs: CREC Ref. No. 2020.311
Record Dates: First submitted 2022-02-28; First posted 2022-03-09 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Fasting
Keywords: Gastric ultrasound; Gastric emptying
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Gastric ultrasound — Gastric ultrasound upon fasting, after 4 hours, and after nasogastric aspiration, to estimate gastric volume

SUMMARY:
Serial gastric ultrasound assessments to assess the effect of fasting for 4 hours on gastric volume in mechanically ventilated patients in the ICU fasted for extubation.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age,
* mechanically ventilated patients in the ICU,
* intubated with endotracheal
* enteral feeding for over 6 hours before fasting

Exclusion Criteria:

* BMI > 40, pregnant, fine bore nasogastric tube, mechanical obstruction to gastric emptying, history of upper GI surgeries

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated patients in the ICU who had been on enteral feeding via nasogastric tube, fasted for extubation
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Difference in gastric volume before and after 4 hours of fasting | Over 4 hours
  Ultrasound measurement of gastric antrum dimenstions (antero-posterior and cranio-caudal dimensions) before and after 4 hours of fasting

CONTACTS AND LOCATIONS:
Overall Officials: Esther Tang, Principal Investigator — Prince of Wales Hospital, Shatin, Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided